CLINICAL TRIAL: NCT00668603
Title: Comparison of Vascular Findings Between Symptomatic and Asymptomatic Postmenopausal Women Before and During Hormone Therapy: A Randomized, Placebo-controlled Prospective Study
Brief Title: Comparison of Vascular Findings Between Symptomatic and Asymptomatic Postmenopausal Women Before and During Hormone Therapy (HRT)
Acronym: SYMPTOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Päivikki and Sakari Sohlberg Foundation, Finland (Other); Emil Aaltonen Foundation (Other); Finnish Medical Foundation (Network)
Responsible Party: Principal Investigator, Tomi S. Mikkola, Associate Professor, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U1030N1016; HUS-231911
Record Dates: First submitted 2008-04-24; First posted 2008-04-29 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Postmenopausal Vasomotor Symptoms; Cardiovascular Disease
Keywords: Postmenopausal vasomotor symptoms; Hot flush; Vascular function; Cardiac function; Cardiovascular risk factor
MeSH Terms: conditions — Cardiovascular Diseases; Hot Flashes | interventions — Estradiol; Gels

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Experimental): Postmenopausal women with severe vasomotor symptoms
  Interventions: Drug: 17-b-estradiol; Drug: 17-b-estradiol + medroxyprogeterone acetate; Drug: 17-b-estradiol hemihydrate; Drug: placebo pill + gel
- 1 (Experimental): Postmenopausal women without vasomotor symptoms
  Interventions: Drug: 17-b-estradiol; Drug: 17-b-estradiol + medroxyprogeterone acetate; Drug: 17-b-estradiol hemihydrate; Drug: placebo pill + gel

INTERVENTIONS:
Drug: 17-b-estradiol — 2mg oral daily for 6 months
Drug: 17-b-estradiol + medroxyprogeterone acetate — 2mg E2 + 5mg MPA daily for 6 months
  Other Names: Indivina
Drug: 17-b-estradiol hemihydrate — 1 mg skin gel daily for 6 months
  Other Names: Divigel
Drug: placebo pill + gel — placebo daily for 6 months

SUMMARY:
Recent large randomized, placebo-controlled studies assessing the health effects of HT question the overall benefits of long term HT, especially with respect to cardiovascular disease. However, recently menopausal women with severe hot flushes were mostly excluded from these trials. This was unfortunate since vasomotor symptoms may reflect different vascular sensitivity to estrogen or its deficiency, and therefore, the vascular responses to HT in women with and without hot flushes can differ.

Aims of the present project are

1. to compare vascular, cardiac and sympathetic function in recently menopausal women with or without severe vasomotor symptoms
2. in a randomized placebo controlled clinical trial investigate vascular response to oral and trans-dermal HT.

DETAILED DESCRIPTION:
We recruit 160 healthy postmenopausal women between ages 48-55. Eighty women must have severe vasomotor symptoms (at least seven severe or moderate hot flush attacks per day) whereas 80 comparators must be symptomless (no hot flushes). Thorough vascular function and risk factor assessments will be done, including clinical assessment of autonomic nervous system, endothelial function measurements, 24-hour ECG and blood pressure evaluation, and lipid and various other vascular surrogate marker measurements. In the first part of the study we compare these baseline measurements between women with or without severe vasomotor symptoms. In the second part of the study the women are randomized to receive placebo, oral estrogen, oral estrogen plus progestin or transdermal estrogen for 6 months. After the treatments the baseline assessments are repeated.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women between ages 48-55
* Minimum of 6 months and maximum of 36 months from last menstrual period
* Postmenopausal status of these women will be confirmed by level of FSH that should exceed 30 U/l
* Eighty women must have severe vasomotor symptoms (at least seven severe or moderate hot flush attacks per day) whereas eighty comparators must be symptomless

Exclusion Criteria:

* smoking
* hysterectomy
* dyslipidemia
* overt hypertension (blood pressure > 140/90)
* diabetes
* any regular medication
* HT in the previous 3 months
* body mass index over 27

Ages: 48 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2005-08; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Vascular function | 0 and 6 months

SECONDARY OUTCOMES:
Cardiac and sympathetic function | 0 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tomi S Mikkola, MD, Principal Investigator — Associate Professor
Locations (1):
- Helsinki University Hospital, Department of Obstetrics and Gynecology, Helsinki, Helsinki, Finland

REFERENCES:
- [Background] Mikkola TS, Clarkson TB. Estrogen replacement therapy, atherosclerosis, and vascular function. Cardiovasc Res. 2002 Feb 15;53(3):605-19. doi: 10.1016/s0008-6363(01)00466-7. PMID 11861031
- [Background] Mikkola TS, Clarkson TB. Coronary heart disease and postmenopausal hormone therapy: conundrum explained by timing? J Womens Health (Larchmt). 2006 Jan-Feb;15(1):51-3. doi: 10.1089/jwh.2006.15.51. No abstract available. PMID 16417418
- [Background] Collins P, Rosano G, Casey C, Daly C, Gambacciani M, Hadji P, Kaaja R, Mikkola T, Palacios S, Preston R, Simon T, Stevenson J, Stramba-Badiale M. Management of cardiovascular risk in the peri-menopausal woman: a consensus statement of European cardiologists and gynaecologists. Eur Heart J. 2007 Aug;28(16):2028-40. doi: 10.1093/eurheartj/ehm296. Epub 2007 Jul 20. PMID 17644507
- [Derived] Tuomikoski P, Mikkola TS, Tikkanen MJ, Ylikorkala O. Hot flushes and biochemical markers for cardiovascular disease: a randomized trial on hormone therapy. Climacteric. 2010 Oct;13(5):457-66. doi: 10.3109/13697131003624656. PMID 20443719
- [Derived] Tuomikoski P, Ebert P, Groop PH, Haapalahti P, Hautamaki H, Ronnback M, Ylikorkala O, Mikkola TS. Effect of hot flushes on vascular function: a randomized controlled trial. Obstet Gynecol. 2009 Oct;114(4):777-785. doi: 10.1097/AOG.0b013e3181b6f268. PMID 19888035
- [Derived] Tuomikoski P, Ebert P, Groop PH, Haapalahti P, Hautamaki H, Ronnback M, Ylikorkala O, Mikkola TS. Evidence for a role of hot flushes in vascular function in recently postmenopausal women. Obstet Gynecol. 2009 Apr;113(4):902-908. doi: 10.1097/AOG.0b013e31819cac04. PMID 19305337